CLINICAL TRIAL: NCT06065228
Title: Development of a Therapeutic Endpoint in Pediatric IBD Conditions
Brief Title: Therapeutic Endpoint in Pediatric IBD Conditions
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Julia Finkel, Professor of Anesthesiology and Pediatrics, Children's National Research Institute
Other Study IDs: STUDY00000658
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- UC
  Interventions: Other: AlgometRx Nociometer
- CD
  Interventions: Other: AlgometRx Nociometer

INTERVENTIONS:
Other: AlgometRx Nociometer — Physiologic characterization of disease activity

SUMMARY:
The purpose of this clinical study is the development of physiologic endpoint of inflammation in pediatric patients diagnosed with inflammatory bowel disease (IBD), specifically subtypes Crohn's disease (CD) and ulcerative colitis (UC). The novel medical device evaluates the patient's sensory response to each of the three sensory nerve fiber types. Data from the device provides an assessment of disease activity and a more precise approach to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 6 years of age at screening.
* Documentation of an IBD diagnosis as evidenced by history

Exclusion Criteria:

* Documented history of eye disease precluding pupillometry
* Patients who are unwilling or unable to participate due to developmental delays or ongoing psychological diagnoses.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study proposes to enroll patients diagnosed with IBD in a longitudinal design.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is the measurement of the nociceptive index for clinical output. | 1 Year

SECONDARY OUTCOMES:
The secondary objective of this study is the characterization of the nociceptive index in IBD populations in response to standard of care interventions. | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided